CLINICAL TRIAL: NCT02216175
Title: Phase 2/3 Clinical Trial to Assess the Effect of a Sublingual Treatment Phase Prior to Oral Immunotherapy in Children With Cow's Milk Allergy
Brief Title: Improving the Safety of Oral Immunotherapy for Cow's Milk Allergy
Acronym: SOCMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: JP Moulton Charitable Foundation (Other); Sociedad Española de Alergología e Inmunología (Unknown); Sociedad Española de Inmunología Clínica, Alergología y Asma Pediátrica (Unknown)
Responsible Party: Principal Investigator, Paul Turner, MRC Clinician Scientist, Clinical Senior Lecturer and Hon Consultant in Paediatric Allergy & Immunology, Imperial College London
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18SM4569; 18/LO/1070 (Other: NHS Human Research Authority)
Record Dates: First submitted 2014-08-07; First posted 2014-08-13 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Food Allergy
Keywords: Cow's milk allergy; Desensitisation; Safety
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SLIT followed by Conventional OIT (Experimental): Participants will receive up to 7 months of SLIT followed by 6 months conventional OIT to cow's milk
  Interventions: Other: SLIT to cow's milk; Other: Conventional OIT to cow's milk
- Conventional OIT (Active Comparator): Participants will receive up to 7 months of low dose OIT, followed by 6 months conventional OIT to cow's milk
  Interventions: Other: Low dose OIT; Other: Conventional OIT to cow's milk
- Delayed start OIT (Placebo Comparator): Participants will receive up to 7 months placebo, followed by 6 months conventional OIT to cow's milk
  Interventions: Other: Conventional OIT to cow's milk

INTERVENTIONS:
Other: SLIT to cow's milk — Sublingual immunotherapy
  Arms: SLIT followed by Conventional OIT
Other: Low dose OIT — Oral Immunotherapy (low dose)
  Arms: Conventional OIT
Other: Conventional OIT to cow's milk — Oral Immunotherapy

SUMMARY:
Allergy to cow's milk is the most common food allergy affecting children. There is currently no accepted routine clinical therapy to cure milk allergy. Recently studies have attempted to induce desensitisation using small daily doses of cow's milk, predominantly by the oral route (oral immunotherapy, OIT). Although this therapy works for some people, its effects are not generally long lasting and it is associated with significant side effects during protocol, including potentially life-threatening allergic reactions.

Pilot data suggests that sublingual immunotherapy (SLIT, where allergen is held under the tongue, rather than swallowed) can also induce a degree of desensitisation, but with fewer adverse events. However, the degree of desensitisation induced appears to be lower than that with oral immunotherapy.

The investigators wish to determine whether a sublingual pretreatment phase can improve the safety of conventional OIT in cow's milk allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Allergic to 1.44g CM protein (approx. 40ml fresh milk) or less, at DBPCFC prior to randomisation
2. Informed consent of parent/legal guardian, patient assent where possible

Exclusion Criteria:

1. Required previous admission to an intensive care unit for management of an allergic reaction.
2. Significant symptoms of non---IgE---mediated CM allergy within the previous 12 months.
3. Children with a past history of CM allergy currently consuming CM-containing products other than extensively--heated milk in baked foods (e.g. biscuits, cakes).
4. Poorly controlled asthma within the previous 3 months (as defined by clinician judgement with reference to the ICON consensus), or asthma requiring treatment with >5 days oral corticosteroids within the previous 3 months.
5. Moderate---severe eczema, defined as requiring more than once daily application of 1% hydrocortisone as maintenance treatment despite appropriate use of emollients (eczema is not otherwise an exclusion criteria)
6. Clinically significant chronic illness (other than asthma, rhinitis or eczema)
7. History of symptoms of eosinophilic oesophagitis, irrespective of cause
8. Undergoing specific immunotherapy to another allergen and within the first year of treatment.
9. Receiving anti--IgE therapy, oral immunosuppressants, beta---blocker or ACE inhibitor.
10. Pregnancy
11. Unwilling or unable to fulfil study requirements

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Adverse events in participants | 1 year
  Proportion of participants experiencing adverse events (excluding mild, non-transient symptoms) conventional OIT to cow's milk in phase 2, in those who have received SLIT pretreatment compared to placebo.

SECONDARY OUTCOMES:
Incidence of adverse events | 1 year
  Incidence of adverse events experienced (including rate of withdrawals, and anaphylaxis/adrenaline use during updosing)
Eliciting dose(mg cow's milk protein) at DBPCFC after each phase of immunotherapy | 1 year
  Efficacy defined at Double-blind, placebo-controlled food challenge (DBPCFC) as the proportion of study participants experiencing:
  * No symptoms (or only mild transient symptoms) to 8 grams CM protein (approx. 250mls fresh milk) ("Complete desensitisation")
  * No symptoms (or only mild transient symptoms) to at least 1.4 grams CM protein (approx. 45mls fresh milk) ("Partial desensitisation")
  * At least a 10--fold increase in eliciting dose (defined as the lowest dose which elicits objective symptoms or signs at challenge). …at 6 and 12 months in the different treatment groups
Change in Health-related quality of life (HRQL) from baseline - assessed using FAQLQ - after each phase of immunotherapy | 15 months
  Change in HRQL measures at 6, 12 and 15 months from baseline, as assessed in study participants and their parent/carer using the following validated questionnaire:
  - Food Allergy Quality of Life Questionnaires (FAQLQ)
Change in Health-related quality of life (HRQL) from baseline - assessed using FAIM - after each phase of immunotherapy | 15 months
  Change in HRQL measures at 6, 12 and 15 months from baseline, as assessed in study participants and their parent/carer using the following validated questionnaire:
  - Food Allergy Independent Measure (FAIM)
Change in Health-related quality of life (HRQL) from baseline - assessed using Change in EQ-5D from baseline - after each phase of immunotherapy | 15 months
  Change in HRQL measures at 6, 12 and 15 months from baseline, as assessed in study participants and their parent/carer using the following validated questionnaire:
  - EQ-5D - a standardized instrument for use as a measure of health outcome.
Change in self-efficacy after each phase of immunotherapy | 15 months
  Change in self-efficacy at 6, 12 and 15 months from baseline, as assessed in study participants and their parent/carer using validated questionnaire.
Immunological outcomes | 12 months
  Change in skin prick test wheal (mm), end-point titration skin prick test, allergen-specific IgE (KuA/l) between baseline and post immunotherapy
Immunological outcome: skin prick test | 12 months
  Change in skin prick test wheal (mm) and end-point titration skin prick test between baseline and post immunotherapy
Immunological outcomes: Allergen-specific IgE | 12 months
  Change in allergen-specific IgE (KuA/l) between baseline and post immunotherapy
Peptide microarray | 12 months
  Trend in CM-peptide binding during OIT

CONTACTS AND LOCATIONS:
Locations (2):
- Niño Jesús Hospital, Madrid, Spain
- Imperial College London / Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Turner PJ, Duca B, Chastell SA, Alvarez O, Bazire R, Vazquez-Ortiz M, Rodriguez Del Rio P. IgE-sensitization predicts threshold but not anaphylaxis during oral food challenges to cow's milk. Allergy. 2022 Apr;77(4):1291-1293. doi: 10.1111/all.15195. Epub 2021 Dec 14. No abstract available. PMID 34874567

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT02216175/Prot_SAP_000.pdf